CLINICAL TRIAL: NCT01706952
Title: Comparison of Topical Vasoconstriction in Endoscopic Sinus Surgery: Cocaine Versus Adrenaline
Brief Title: Comparison of Topical Vasoconstriction in Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marc Tewfik (Other)
Responsible Party: Sponsor-Investigator, Marc Tewfik, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12-251-SDR
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Chronic Sinusitis
Keywords: Endoscopic sinus surgery; Bleeding; Topical Vasocontriction; Cocaine; Adrenaline
MeSH Terms: conditions — Hemorrhage | interventions — Cocaine; Epinephrine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cocaine (Experimental): Cocaine 4%. Three cotton neuropatties will be soaked with 4% cocaine. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This intervention will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Interventions: Drug: Cocaine; Drug: Adrenaline
- Adrenaline (Active Comparator): Adrenaline 1/1.000 Three cotton neuropatties will be soaked with Adrenaline 1/1,000. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Interventions: Drug: Cocaine; Drug: Adrenaline

INTERVENTIONS:
Drug: Cocaine — Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Other Names: Brand Name: Cocaine Hydrochloride Sterile Topical Solution; Generic Name: Cocaine Hydrochloride Sterile Topical Solution; Active Ingredients: Cocaine hydrochloride; Concentration: 4%; Code: 1200; Format: 5 x 5 mL; DIN: 01962388; UPC: 057513012006; Preservative: Yes; Special feature: Latex Free Stopper
Drug: Adrenaline — Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
  Other Names: Epinephrine

SUMMARY:
The purpose of our study is to assess the effect of topical vasoconstriction (cocaine 4% versus adrenaline 1/1000) on the surgical field during endoscopic sinus surgery.

DETAILED DESCRIPTION:
Chronic Rhinosinusitis (CRS) is one of the most common chronic illnesses in North America, with an incidence of approximately 13 per cent in the US.

Endoscopic sinus surgery (ESS) has become standard treatment for patients with chronic rhinosinusitis (CRS) unresponsive to maximum medical treatment. The success of surgery depends on several factors, an adequate surgical field is among the most important factors in preventing complications in ESS.

Topical vasoconstrictors, such as adrenaline and cocaine has been widely used. To date no studies exist comparing the use of topical cocaine with adrenaline in ESS.

The purpose of this study is to assess the effect of topical cocaine 4% versus adrenaline on intra-operative bleeding during ESS and to describe the phisiologic changes with the use of topical vasocontrictors. A secondary objective is to describe the phisiologic changes with the use of topical vasocontrictors

Study Design:

A prospective randomized single-blind controlled trial will be conducted. The surgeon performing the ESS and evaluating the bleeding will not be present at the time of injection, and so will remain blinded.

All patients over the age of 18 years undergoing bilateral ESS for chronic sinusitis at McGill University Health Center will be invited to participate. The study will be conducted from November 2012 until the number required of patients is enrolled.

Topical vasoconstriction technique After oral intubation, vital signs and all anaesthetic parameters will be kept as constant as possible for the duration of the surgery. Three cotton neuropatties will be soaked with 4% cocaine. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined. In the other side, three cotton neuropaties will be soaked with adrenaline 1:1000 and placed in the same positions than the others. Then the patient will be draped and both sides will be injected with xylocaine 2% and adrenaline 1:100.000. After this we will wait for 10 minutes and the surgery will be initiated.

At the commencement of surgery and at regular 15-minute intervals, the operating surgeon will estimate the intensity of bleeding in the operative field. The extent of nasal bleeding will be evaluated according to the validated scale used by Boezaart. At each assessment, other parameters including mean arterial blood pressure (MAP), heart rate, and end tidal CO2 will be recorded into a chart by the co-investigator.

The total blood loss will be collected and recorded separately for each side. Separate suction tubes and canisters will be used for each side. The total blood loss will be measured by subtracting the amount of saline solution used to rinse the surgical field from the amount of blood and fluids suctioned from the surgical field. Although this method of estimating the intra operative blood loss is not flawless as some blood and fluids usually fall posteriorly into the nasopharynx and are later suctioned by the anesthesiologist prior to extubation, this amount is deemed to be negligible.

Proposed data analysis: The data will be collected by the co-investigator. Patient names and other specific identifiers will not be included. Data will be entered into an Excel spreadsheet and statistical analysis will be applied with SPSS vs.13.

ELIGIBILITY:
Inclusion Criteria:

- Patients older than 18 years undergoing bilateral ESS for chronic sinusitis.

Exclusion Criteria:

* Patients with heart disease
* History of bleeding diathesis
* Patients with untreated or poorly controlled high blood pressure
* Aspirin, anticoagulant or natural herbal medication usage in the last 4 weeks
* Hypersensitivity to adrenaline or cocaine
* Significant asymmetry between the right and left side disease extent as determine by findings on their pre-operative CT scan and nasal endoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Tewfik, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Constanza J Valdes, MD, Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre; Mark Samaha, MD, Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Department of Otolaryngology-Head and Neck Surgery. McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Result] Valdes CJ, Bogado M, Rammal A, Samaha M, Tewfik MA. Topical cocaine vs adrenaline in endoscopic sinus surgery: a blinded randomized controlled study. Int Forum Allergy Rhinol. 2014 Aug;4(8):646-50. doi: 10.1002/alr.21325. Epub 2014 Mar 26. PMID 24678064

RESULTS

PARTICIPANT FLOW:
Groups:
- Cocaine/Adrenaline: Cocaine: Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Adrenaline: Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
  Three cotton neuropatties will be placed in each side of the nostril. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This intervention will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
Period: Overall Study
Arm/Group | Cocaine/Adrenaline
Started | 45
Completed | 37
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: 23 were male, 14 were female
Groups:
- Cocaine/Adrenaline: Three cotton neuropatties will be placed in each nostril. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This intervention will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Cocaine: Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Adrenaline: Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
Arm/Group | Cocaine/Adrenaline
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.92 (16.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23
Region of Enrollment [Number; unit: participants]
  Canada | 37

OUTCOME MEASURES:

1. Primary Outcome: To Estimate the Change in Bleeding Category (Surgical Field Improvement) as Measured on a Six-point Scale, Measured From 0 (Best Case) to 5 (Worst Case).
Description: 0 No bleeding.
  1. Slight bleeding - no suctioning of blood required.
  2. Slight bleeding - occasional suctioning required. Surgical field not threatened.
  3. Slight bleeding - frequent suctioning required. Bleeding threatens surgical field a few seconds after suction is removed.
  4. Moderate bleeding - frequent suctioning required. Bleeding threatens surgical field directly after suction is removed.
  5. Severe bleeding - constant suctioning required. Bleeding appears faster than can be removed by suction. Surgical field severely threatened and surgery not possible.
  For the primary objective of surgical field grade, we calculated the mean within sides treated with cocaine vs adrenaline and assessed its difference
Time Frame: Every 15 minutes until 300 minutes
Population: EACH SIDE WAS EVALUATED SEPARATELY
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cocaine SIDE: Cocaine 4%. Three cotton neuropatties will be soaked with 4% cocaine. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This intervention will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Cocaine: Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Adrenaline: Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
- Adrenaline SIDE: Adrenaline 1/1.000 Three cotton neuropatties will be soaked with Adrenaline 1/1,000. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Cocaine: Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Adrenaline: Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
Arm/Group | Cocaine SIDE | Adrenaline SIDE
Number analyzed (Participants) | 37 | 37
units on a scale | 2.17 (0.70) | 2.04 (0.75)
Statistical Analysis 1: Comparison: Cocaine SIDE vs Adrenaline SIDE; Data analysis was performed using SPSS version 13 for Windows (SPSS Inc, Chicago, IL). A power study was per formed with a power of 80% and a clinically significant difference in bleeding between the sides of 20% with a significance level of 5% (p < 0.05); Test type: Superiority or Other — For surgical field grade, we calculated the mean within sides and assessed its difference, reporting a 95% confidence interval as calculated by a Student t test. We used the average per patient over time; p = 0.05, t-test, 2 sided; For the primary objective of surgical field grade, we calculated the mean within sides treated with cocaine vs adrenaline and assessed its difference, reporting a 95% con- fidence interval as calculated by a Student t test. As all of these values were measured over time, we used the average per patient over time. The total blood loss per side within subjects was also calculated, with 95% confidence interval again calculated by a Student t test. Once again, we took the average per patient over time as the main outcome. Finally, we used a linear regression with surgical field improvement as the outcome and HR, MAP, or etCO2 as covariates, to investigate which variables may be related to the outcome. As these measures were taken over time, we used repeated measures analysis to investigate how these items correlate over time. In addition to the operating surgeon, the statistician was blinded to the vasoconstrictor allocation

2. Secondary Outcome: Heart Rate
Description: The heart rate (heart beats for minutes) will be recorded every 15 minutes, until the surgery is over or until 300 minutes.
  The Co-investigator will record this data in a special data sheeet For the secondary objective of Heart rate, we calculated the average within sides treated with cocaine vs adrenaline and assessed its difference
Time Frame: Every 15 minutes until 300 minutes
Measure: Mean (Standard Deviation); unit: Heart Beats per minute
Arm/Group | Cocaine SIDE | Adrenaline SIDE
Number analyzed (Participants) | 37 | 37
Heart Beats per minute | 74.68 (13.64) | 73.62 (14.23)

3. Secondary Outcome: Blood Pressure
Description: The mean blood pressure, defined as the average arterial pressure during a single cardiac cycle, will be recorded every 15 minutes, until the surgery is over or until 300 minutes.
  For the secondary objective of blood pressure, we calculated the mean within sides treated with cocaine vs adrenaline and assessed its difference
Time Frame: Every 15 minutes or until 300 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cocaine SIDE | Adrenaline SIDE
Number analyzed (Participants) | 37 | 37
mmHg | 68.02 (11.94) | 68.41 (9.15)

4. Secondary Outcome: End Tidal CO2
Description: The concentration of carbon dioxide (CO2) in the respiratory gases will be recorded every 15 minutes or until 300 minutes.
  For the secondary objective of concentration of carbon dioxide, we calculated the mean within sides treated with cocaine vs adrenaline and assessed its difference
Time Frame: Every 15 minutes or until 300 minutes
Measure: Mean (Standard Deviation); unit: Percentage of carbon dioxide
Arm/Group | Cocaine SIDE | Adrenaline SIDE
Number analyzed (Participants) | 37 | 37
Percentage of carbon dioxide | 32.26 (3.24) | 31.69 (2.83)

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of hospital stay, an average of 8 hours, maximum stay up to 24 hours.
Groups:
- Cocaine: Cocaine 4%. Three cotton neuropatties will be soaked with 4% cocaine. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This intervention will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Cocaine: Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Adrenaline: Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
- Adrenaline: Adrenaline 1/1.000 Three cotton neuropatties will be soaked with Adrenaline 1/1,000. One neuropattie will be placed in the sphenoethmoidal recess, one in the middle meatus, and one in the anterior end of the middle turbinates on the side that the randomization has determined.
  This will be done before the beginning of the surgery, and will be left in the nose for 10 minutes, this will be done just once. After the 10 minutes, the neuropatties will be taken out of the nose.
  Cocaine: Pledgets soaked in 4% cocaine hydrochloride solution were placed intranasally (one side).
  Adrenaline: Pledgets soaked in 1/1000 adrenaline solution were placed intranasally (one side).
Arm/Group | Cocaine | Adrenaline
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No